CLINICAL TRIAL: NCT06926049
Title: The Effect of The Mindfulness-Based Psycho-Educational Program Focused on Emotions on Difficulties in Emotion Regulation, Depressive Symptoms and Hope Level in Schizophrenia Patients
Brief Title: The Mindfulness-Based Psycho-Educational Program Focused on Emotion Regulation Strategies
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Figen Şengün İnan, ASSOCIATE PROFESSOR DOCTOR, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Figen ŞENGÜN İNAN
Record Dates: First submitted 2025-04-07; First posted 2025-04-13 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Depressive Symptoms; Hope; Difficulties of Emotion Regulation
Keywords: difficulties of emotion regulation; depressive semptoms; hope; Psychiatric nursing
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: In the study, 48 schizophrenia patients were taken as sampling, 24 of which were experimental and 24 were control.
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the study, it is not possible to blind the researcher implementing the intervention and the participants. To prevent bias in the study, the pretest will be applied before randomization. It is planned to blind the statistical and report writing process in the study. The assignment of schizophrenia patients to the intervention and control groups will be made by a statistician independent of the study. The researcher and schizophrenia patients will not know which group they are in until the application begins. After applying the follow-up tests, the researcher will code the data as A and B groups and transfer it to SPSS. With this method, it is planned that the statistician will do the analysis and reporting without knowing which group is the intervention and which group is the control group. It is planned to explain the codes of the groups after the analysis and reporting of the data. In this way, detection bias, statistical bias, and reporting bias will be prevented
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental: The Effect of The Mindfulness-Based Psycho-Educational Program Focused on Emotions (Experimental): The mindfullness based psychoeducation program focusing on emotions to be carried out with the experimental group is planned as 5 sessions. The sessions are planned to be held in 2 groups of 12 people each. The duration of a session is planned as 45-60 minutes. Group psychoeducation with the experimental group will be carried out face to face every week. The appropriate day for the sessions will be decided with the members of each group. The same group session will be held on the same day and time every week.
  Interventions: Other: The Effect of The Mindfulness-Based Psycho-Educational Program Focused on Emotions
- no intervention (No Intervention): Waiting list group after the follow-up tests were completed, it was planned to apply the 5-session group psychoeducation applied to the intervention group in the same way to the control group, upon their request.

INTERVENTIONS:
Other: The Effect of The Mindfulness-Based Psycho-Educational Program Focused on Emotions — The mindfulness based psychoeducation program focusing on emotions that aims to reduce the difficulties in regulating emotions and depressive symptoms in schizophrenia patients and to increase the level of hope.
  Arms: Experimental: The Effect of The Mindfulness-Based Psycho-Educational Program Focused on Emotions

SUMMARY:
In this study, the effects of a mindfulness-based emotion-focused psychoeducation program applied to individuals diagnosed with schizophrenia on emotion regulation difficulties, depressive symptoms, and hope levels will be examined. The research will be carried out as a randomized controlled experimental study with a pre-test-post-test and follow-up design.

DETAILED DESCRIPTION:
Schizophrenia is a chronic illness that begins at a young age and leads to impairments in thought, perception, and affect. Patients experience a loss of functionality in occupational, social, and personal areas and face emotional challenges such as depression, anxiety, and hopelessness. Difficulties in emotion regulation are common among individuals with schizophrenia, making disease management more challenging.

Emotion regulation refers to the process of recognizing, accepting, and managing emotions using appropriate strategies. Literature indicates that difficulties in emotion regulation among individuals with schizophrenia are associated with depression and an increased risk of suicide. Mindfulness-based interventions have been found effective in enhancing emotion regulation skills and reducing depressive symptoms, rumination, and hallucinations.

This study aims to examine the effects of a mindfulness-based psychoeducation program for individuals diagnosed with schizophrenia on emotion regulation difficulties, depressive symptoms, and levels of hope. The findings are expected to contribute to nurse-led interventions that support the mental health and rehabilitation process of patients.

ELIGIBILITY:
Inclusion Criteria:

1. Being diagnosed with schizophrenia according to DSM-5 diagnostic criteria
2. Being between 18-65 years old
3. Not having any problems with communication
4. Being literate
5. Being willing to participate in the research
6. Having schizophrenia for at least 2 years

Exclusion Criteria:

1. Having a neurological disease
2. Having a neurocognitive disease
3. Having comorbid depression according to DSM-5 diagnostic criteria
4. Being a substance abuser
5. Having participated in and currently receiving a structured psychotherapeutic intervention program within the last year

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Difficulties in Emotion Regulation Scale-Brief Form (DERS-16) | Change from baseline in the mean emotion regulation difficulties scores at the 1st-month follow-up and the 3rd-month follow-up. (baseline, 1st month follow-up, 3rd month follow-up)
  The scale is a 16-item self-report measure, developed by Bjureberg et al. (2016). DERS-16 is used to evaluate various aspects of emotion regulation difficulties. It comprises five subscales, namely Clarity (e.g., "I have difficulty making sense of my feelings"), Goals (e.g., "When I'm upset, I have difficulty getting work done"), Impulse (e.g., "When I'm upset, I feel out of control"), Strategies (e.g., "When I'm upset, I start to feel very bad about myself"), and Non-acceptance (e.g., "When I'm upset, I feel like I am weak"). The items in DERS-16 are rated on a 5-point Likert scale ranging from 1 (almost never) to 5 (almost always). Higher scores indicate greater emotion dysregulation. There are no reverse-coded items in the scale.

SECONDARY OUTCOMES:
Beck Depression Inventory (BDI) | Change from baseline in the mean depression scores at the 1st-month follow-up and the 3rd-month follow-up. (baseline, 1st month follow-up, 3rd month follow-up)
  It was developed by Beck and his colleagues to control the presence and severity of depression. The scale consists of 21 items. The items consist of four items that define a specific behavioral pattern and are scored from zero to three. The score that can be obtained from the scale varies between 0-63. The aim of the scale is to express the symptoms of depression in numbers rather than to diagnose any depression in the participants. It was determined that the presence and severity of depression is higher as the total score increases. Minimal depression will be determined between 0-9 points, Mild depression 10-16 points, Moderate depression 17-29 points and Severe depression 30-63 points. It measures the physical, emotional and cognitive symptoms seen in depression. The higher the total score, the more severe the depression.
Schizophrenia Hope Scale (SHS) | Change from baseline in the mean hope score at the 1st-month follow-up and the 3rd-month follow-up. (baseline, 1st month follow-up, 3rd month follow-up)
  It is a scale developed by Choe (2014) to determine the hope levels of individuals diagnosed with schizophrenia. The scale, which consists of a total of 9 questions, is a three-point Likert type (0=disagree, 1=agree 2=strongly agree). The total score obtained from the scale is between 0 and 18. The scale does not have a cut-off point, and high scores obtained from the scale are interpreted as individuals diagnosed with schizophrenia having high levels of hope.

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University, Ankara, Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] O'Driscoll C, Laing J, Mason O. Cognitive emotion regulation strategies, alexithymia and dissociation in schizophrenia, a review and meta-analysis. Clin Psychol Rev. 2014 Aug;34(6):482-95. doi: 10.1016/j.cpr.2014.07.002. Epub 2014 Jul 24. PMID 25105273
- [Background] Ludwig L, Werner D, Lincoln TM. The relevance of cognitive emotion regulation to psychotic symptoms - A systematic review and meta-analysis. Clin Psychol Rev. 2019 Aug;72:101746. doi: 10.1016/j.cpr.2019.101746. Epub 2019 Jun 14. PMID 31302506
- [Background] Lawlor C, Hepworth C, Smallwood J, Carter B, Jolley S. Self-reported emotion regulation difficulties in people with psychosis compared with non-clinical controls: A systematic literature review. Clin Psychol Psychother. 2020 Mar;27(2):107-135. doi: 10.1002/cpp.2408. Epub 2020 Feb 12. PMID 31661593
- [Background] Hawton K, Sutton L, Haw C, Sinclair J, Deeks JJ. Schizophrenia and suicide: systematic review of risk factors. Br J Psychiatry. 2005 Jul;187:9-20. doi: 10.1192/bjp.187.1.9. PMID 15994566
- [Background] Gratz, K.L., Roemer, L. (2004). Multidimensional Assessment of Emotion Regulation and Dysregulation: Development, Factor Structure, and Initial Validation of the Difficulties in Emotion Regulation Scale. Journal of Psychopathology and Behavioral Assessment 26, 41-54. https://doi.org/10.1023/B:JOBA.0000007455.08539.94
- [Background] Cho M, Jang SJ. Effect of an emotion management programme for patients with schizophrenia: A quasi-experimental design. Int J Ment Health Nurs. 2019 Apr;28(2):592-604. doi: 10.1111/inm.12565. Epub 2018 Dec 25. PMID 30585413